CLINICAL TRIAL: NCT06485726
Title: Valproate Versus Propranolol in Migraine, a Randomized Controlled Trial
Brief Title: Valproate Versus Propranolol in Migraine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01012019
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Migraine Disorders
Keywords: propranolol; valproate; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid; Propranolol

STUDY DESIGN:
Intervention Model Description: We will assess The number of migraine days after three months of treatment and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. Treatment safety was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; participants received either lacosamide or propranolol from a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 600 labels for each drug labelled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 600. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrollment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included valproate, and Drug B included propranolol. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- valproate arm (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive valproate 500-1000 mg daily for three months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. Treatment safety was evaluated by monitoring and documenting patients' treatment-emergent adverse events (TEAE) through regular follow-up procedures for three months.
  Interventions: Drug: Valproic Acid 500 MG
- Propranolol group (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive propranolol 160 mg once daily for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of lacosamide was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Valproic Acid 500 MG — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The treatment safety was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group A
  Arms: valproate arm
Drug: Propranolol — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The treatment safety was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group B
  Arms: Propranolol group

SUMMARY:
Investigators aim to compare the effect of valproate versus propranolol in migraine by assessing the absolute reduction in MMD in each group and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency.

DETAILED DESCRIPTION:
Investigators will enrol 600 migraine patients who are diagnosed according to ICHD3-beta criteria in our study and will use a questionnaire to detect their demographic and clinical features (disease duration, attack frequency, and duration, pain intensity assessed by the visual analogic scale and we have two groups the first group will include 300 patients and will receive 500-1000 mg valproate daily, and the second group will receive propranolol 160 mg per day. Investigators will assess The number of migraine days after three months of treatment and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency. The safety of lacosamide was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.

ELIGIBILITY:
Inclusion Criteria:

Naive migraine patients, according to the International Classification of Headache Disorders 3rd edition, aged 18-75 years,

Exclusion Criteria:

* Patients with major neurological disorders such as (epilepsy, ischemic or hemorrhagic stroke, multiple sclerosis, mitochondrial diseases, brain tumours, and patients with essential tremors.
* Patients with major systemic diseases such as malignancy, collagen, liver, and renal diseases.
* Patients with cardiovascular diseases like hypertension (systolic blood pressure of more than 130 and/or diastolic blood pressure of more than 85 mm/Hg on at least three different occasions, diabetes (fasting plasma glucose level >126 mg/dl and/or a casual plasma glucose >200 mg/dl and/or HbA1C more than 6.5.
* patients with valvular and ischemic heart diseases, bradycardia or heart blocks, congestive heart failure
* patients who received prophylactic treatment for migraine,
* patients with any contraindications to drugs used in the study
* patients with bronchial asthma, chronic obstructive pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
The change in migraine days per 28 days | 28 days
  The investigators will assess the change in migraine days per 28 days in each group.

SECONDARY OUTCOMES:
The total number of migraine days after three months of treatment | 3 months
  The investigators will assess the total migraine days after three months of regular use of 500-1000 mg valproate daily or propranolol (160 mg once daily).
The percentage of patients who achieved ≥ 50% change in the monthly migraine days frequency compared to the baseline frequency. | 3 months
  We will assess The percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency in each group
HIT-6 score absolute change in each group after three months of treatment | 3 months
  The investigators assessed the absolute change in HIT6 score; the Headache Impact Test-6 (HIT-6) evaluated the burden of headache in each group; the HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress, the patient answers each of the six related questions using one of the following five responses: "never," "rarely," "sometimes," "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a more significant impact of headaches on the daily life of the respondent. It has four impact grades: little-to-no impact (HIT-6 score: 36-49), moderate impact (HIT-6 score: 50-55), substantial impact (HIT-6 score: 56-59), and severe impact (HIT-6 score: 60-78)
Incidence of Treatment-Emergent Adverse Events | 3 months
  The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
The principal investigator, Mohamed G. Zeinhom, may provide all the data supporting this research's findings upon reasonable request.

REFERENCES:
- [Result] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523
- [Result] Mushet GR, Miller D, Clements B, Pait G, Gutterman DL. Impact of sumatriptan on workplace productivity, nonwork activities, and health-related quality of life among hospital employees with migraine. Headache. 1996 Mar;36(3):137-43. doi: 10.1046/j.1526-4610.1996.3603137.x. PMID 8984084